CLINICAL TRIAL: NCT04768933
Title: Parental Notions and Clinical Experiences About Child's Gut Comfort, Overall Satisfaction and Sense of Well-being When Consuming a New Toddler Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20.14.INF
Record Dates: First submitted 2020-12-17; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Digestion; Happiness; Temperament
Keywords: prebiotic; digestion; child development; temperament

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toddler Milk Group (Experimental): All enrolled subjects with be provided a new toddler milk for 28 days. Aligned with clinical and label recommendations, they will be required to intake at least 3 servings of 130 ml per day.
  Interventions: Dietary Supplement: Toddler Milk

INTERVENTIONS:
Dietary Supplement: Toddler Milk — At least three 130 mL servings daily of study formula are recommended for a total daily intake of 390 mL. Study participants will continue this feeding regimen Days 4 to 28 (approximately 4 weeks).

SUMMARY:
This is a prospective, open-label, single-arm study in a real-world setting of healthy Chinese toddlers provided with new toddler milk for a total of 4 weeks (28 days).

DETAILED DESCRIPTION:
The new toddler milk contains prebiotic and an optimized fat blend of bovine milk fat, vegetable fats, and a LC-PUFA oil mixture (providing DHA and ARA). The prebiotic and bovine milk fat-based blend have shown to be able to improve digestive comfort and milk taste. Physiological factors such as physical discomfort has been shown to be associated with negative emotionality and temperament (Putnam 2012). Therefore, the investigators hypothesize that by improving digestive comfort, they are able to influence child temperament, happiness, and other behavioral characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy toddlers born at term (37-42 weeks of gestation).
2. At enrolment visit, toddler age 12-33 months.
3. Birth weight ≥ 2500g and ≤ 4500g.
4. No known milk intolerance / allergies to cow's milk protein.
5. Habitually consuming some cow's milk or other traditional milks.

Exclusion Criteria:

1. Toddler is currently breastfed or is consuming breast milk.
2. Toddler who is experiencing growth faltering (defined as weight for length z score ≤-1.67).
3. History of preterm birth
4. Currently experiencing severe constipation.
5. Currently diagnosed with other Functional Gastrointestinal Disorders.
6. Toddlers who have known cognitive and developmental disorders.
7. Toddlers who are currently participating in or have participated in another clinical trial within 4 weeks prior to trial start.

Ages: 12 Months to 33 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-10-11 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Digestive tolerance | Baseline (week 0) and week 4 (Day 28±2)
  Change in overall digestive tolerance composite scores measured by the Toddler Gut Comfort Questionnaire consisting of 10 questions on parent perceptions of constipation, diarrhea, gassiness, abdominal pain, bloating and other GI-related behaviors.

SECONDARY OUTCOMES:
Temperament | from baseline (week 0) to week 4 (Day 28±2)
  Change in temperament surgency scores derived from the Children's Behavior Questionnaire (CBQ), short version
Child's emotional expressions | at weeks 0 (baseline), 1 (Day 7±2), 2 (Day 14±2), and 4 (Day 28±2).
  Child's emotional expressions such as Happy, Smiling, Surprised, Anger, and Disgust derived from the Anura phone app. In addition, parents will report child's mood including being happy, relaxed and smiling in the Mood Diary.
Milk Satisfaction | at weeks 0 (baseline), 1 (Day 7±2) and 4 (Day 28±2).
  Milk Satisfaction derived from a toddler and parent-reported brief (9-items) Milk Satisfaction Questionnaire The questionnaire consists of questions regarding taste, sweetness, milky taste, nutritional profile, and convenience.
Weight in kilograms | at week 0 (baseline) and week 4 (Day 28±2)
  Weight (kg) will be taken for the purpose of assessing child's growth
Height in centimeters | at week 0 (baseline) and week 4 (Day 28±2)
  Height (cm) will be taken for the purpose of assessing child's growth
Milk intake | at baseline and prospectively during transition period (Day 1-3) and for three consecutive days on week 1 (Day 7±2), 2 (Day 14±2) and 4 (Day 28±2).
  based on 24-hour recall of dairy and non-dairy intake obtained from the Milk Intake Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Information Technology co., LTD, Shanghai, China

IPD SHARING:
Plan to Share IPD: No